CLINICAL TRIAL: NCT03235973
Title: Cladribine Dose Escalation in Conditioning Regimen Prior to Allo-HSCT for Refractory Acute Leukemia and Myelodysplastic Syndromes
Acronym: CEREAL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEREAL-IPC 2016-010
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoblastic, Acute
Keywords: refractory acute leukemia; refractory myelodysplastic syndrome; cladribine dose escalation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine-Cladribine-Busulfan conditioning regimen (Experimental)
  Interventions: Drug: Fludarabine-Cladribine-Busulfan conditioning regimen

INTERVENTIONS:
Drug: Fludarabine-Cladribine-Busulfan conditioning regimen — Conditioning regimen will be performed from day -6 to day -2 and contains:
  * Fludarabine 10 mg/m²/d during 5 days (day-6 to day-2).
  * Cladribine during 5 days (day-6 to day-2) at one the following define dose level:
    * Dose 1: 10 mg/m²/d
    * Dose 2: 15 mg/m²/d
    * Dose 3: 20 mg/m²/d
    * Dose 4: 25 mg/m²/d
  * IV busulfan will be given on day-6 using fixed dose as following:
    * If age ≤ 60 years: starting dose of 130 mg/m²
    * If age > 60 years: starting dose of 100 mg/m² No busulfan will be administered at day-5, allowing the pharmacokinetic (PK) analyses . Subsequent infusion of IV busulfan will be performed from day-4 to day-2 at the dose recommended by PK analyses

SUMMARY:
The investigators focused on patients with refractory acute leukemia or MDS and designed a phase 1 trial of escalated cladribine doses in the Cla-Flu-Bu RTC regimen using PK-guided myeloablative busulfan doses. This scheme allows combining different optimization of RTC experienced over years (Flu-Bu RTC, PK-guided myeloablative busulfan doses, a second purine analog cladribine) to approach a specific platform to treat refractory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* ECOG 0 or 1
* Acute leukemia (AML or ALL) without criteria for CR or high risk MDS without criteria for CR
* Availability of a donor among following oHLA identical sibling oHaploidentical donor o10/10 or 9/10 allele-level HLA matched unrelated donor
* Signed informed consent
* Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen

Exclusion Criteria:

* Contraindication for Allo-HSCT
* Cord blood Allo-HSCT
* Current active disease or positive serology for HIV, and/or HCV with detectable viremia and/ or HBV with positive Hbs Antigen.
* Renal failure with creatinine clearance < 30 ml/ min
* Decompensated haemolytic anaemia
* Hypersensitivity to an active substance or to any of the excipients
* Acute urinary infection
* Pre-existing haemorrhagic cystitis
* Woman of childbearing potential not using an effective contraception .
* Pregnant or lactating women
* Any serious concurrent uncontrolled medical disorder
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-04-28 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
estimation of the maximal tolerable dose,if any,and recommended phase II dose of cladribine administered as in combination with fludarabine and PK-guided IV busulfan prior Allo-HSCT for refractory acute leukemia and myelodysplastic syndrome (MDS) | 30 days after Allo-HSCT
  Occurrence ratio of dose-limiting toxicity defined as any grade ≥ 3 toxicity according to CTCAE (version 4.03 ) attributable to conditioning regimen (extra-medullary toxicity), considered to be related or probably related to the Cla-Fu-Bu RTC by the investigator.

SECONDARY OUTCOMES:
Cumulative incidence of acute Graft versus host disease | 100 days
  Cumulative incidence of acute Graft versus host disease according to Gluckberg's classification
Cumulative incidence of chronic Graft versus host disease | 1 year
  Cumulative incidence of chronic Graft versus host disease according to NIH classification
Cumulative incidence of relapse | 1 year
  Cumulative incidence of relapse at 1 year
Cumulative incidence of Non Relapse Mortality | 100 days, 1 year
  Cumulative incidence of Non Relapse Mortality at day +100 and 1 year after Allo-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Raynier Devillier, MD,PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône, France